CLINICAL TRIAL: NCT03628326
Title: Is Pulmonary Segmentectomy an Anatomical Resection? Evaluation of Visceral Pleural Lumbar Lymphatic Drainage - Anatomo-clinical Correlation.
Brief Title: Evaluation of Visceral Pleural Lumbar Lymphatic Drainage
Acronym: SEGPUL
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: RNI2016-01
Record Dates: First submitted 2018-07-31; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Pulmonary Artery Stenosis
Keywords: Pulmonary artery; 3D reconstruction; Video-assisted thoracic surgery lobectomy; CT angiography; Anatomic variation
MeSH Terms: conditions — Stenosis, Pulmonary Artery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- right lung resection: The investigators sought to identify anatomic variations of the pulmonary arterial tree and assess their respective frequencies.
  Interventions: Other: Pulmonary arterial tree
- left lung resection: The investigators sought to identify anatomic variations of the pulmonary arterial tree and assess their respective frequencies.
  Interventions: Other: Pulmonary arterial tree

INTERVENTIONS:
Other: Pulmonary arterial tree — The investigators performed 3D reconstruction of the pulmonary arterial tree on the CT angiography data set acquired during preoperative work-up.

SUMMARY:
Anatomic variations of the pulmonary arterial tree can cause technical difficulties during pulmonary lobectomy in general and video-assisted thoracic surgery (VATS). Using CT angiography and 3D reconstruction, the investigators sought to identify anatomic variations of the pulmonary arterial tree and assess their respective frequencies.

DETAILED DESCRIPTION:
Purpose Anatomic variations of the pulmonary arterial tree can cause technical difficulties during pulmonary lobectomy in general and video-assisted thoracic surgery (VATS). Using CT angiography and 3D reconstruction, the investigators sought to identify anatomic variations of the pulmonary arterial tree and assess their respective frequencies. Methods the investigators retrospectively studied 88 pulmonary arterial trees in 44 patients having undergone VATS lobectomy for lung cancer over an 18-month period in Amiens University Hospital's Department of Thoracic Surgery. Each CT angiography with 3D reconstruction of the pulmonary arterial tree was performed by two experienced operators, according to a standardized procedure.

ELIGIBILITY:
Inclusion Criteria:

* Any major patient aged 18 years and over who has undergone oncological lung lobectomy for non-small-cell lung cancer located in the thoracic surgery department of the University Hospital of Amiens.
* Nosologic criteria and related to acts: The pathology has already been diagnosed or suspected, and the surgical indication has been validated in the Multidisciplinary Thoracic Oncology Concertation Meeting according to national recommendations.
* These patients will be collected in a database already referenced in the register of the establishment of the University Hospital of Amiens under the reference DRCI T38

Exclusion Criteria:

* Criteria relating to the population:
* Patient under guardianship or curatorship
* Pathology Criteria: Patient with no pulmonary neoplastic disease, patient with locally advanced or metastatic bronchopulmonary cancer
* Criteria relating to the acts: the criteria altering the surgical specimen and thus its anatomical study: patient having had an extemporaneous examination, patient with the antecedents of ipsilateral pulmonary surgery and / or need of decortication

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators studied patients having undergone VATS lobectomy for stage I-II lung cancer at the Amiens University Hospital's Department of Thoracic Surgery between October 2012 and March 2014. We performed 3D reconstruction of the pulmonary arterial tree on the CT angiography data set acquired during preoperative work-up.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Use CT angiography and 3D reconstruction | 18-month
  The primary objective of the present study was to use CT angiography and 3D reconstruction to assess the pulmonary arterial tree and its anatomic variations in patients having undergone VATS lobectomy for stage I-II lung cancer. The investigators studied patients having undergone VATS lobectomy for stage I-II lung cancer at the Amiens University Hospital's Department of Thoracic Surgery between October 2012 and March 2014. The investigators performed 3D reconstruction of the pulmonary arterial tree on the CT angiography data set acquired during preoperative work-up. Patients having undergone CT angiography in another hospital, those not having undergone CT angiography of the arterial tree, and those having been operated on more than once for lung cancer were excluded from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Marçon, MD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No